CLINICAL TRIAL: NCT03656224
Title: Survey of Post-Acute Inpatient Rehabilitation Safety Concerns in the Cancer Population
Brief Title: Survey of Post-Acute Inpatient Rehabilitation Safety Concerns in Participants With Cancer
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2018-0104; NCI-2018-01749 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0104 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-08-27; First posted 2018-09-04 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (survey): Participants complete surveys over 15 minutes at 1-2 days before discharge and at 1 month after discharge.
  Interventions: Other: Survey Administration

INTERVENTIONS:
Other: Survey Administration — Ancillary studies

SUMMARY:
This trial studies a survey of post-acute inpatient rehabilitation safety concerns in participants with cancer. Collecting patients' feedback via surveys may help doctors to learn more about the safety concerns that patients have when they are discharged from the acute inpatient cancer rehabilitation unit.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess patients' perceptions regarding safety after acute inpatient rehabilitation at discharge and after approximately one month from discharge date.

SECONDARY OBJECTIVES:

I. Assess patient's perception of factors impacting continuity of care at discharge and after approximately one month from discharge date.

II. Determine the frequency of reported falls and the circumstance surrounding reported falls during hospitalization and within approximately one month from discharge date.

III. Determine the frequency of reported near falls and the circumstance surrounding reported near falls within approximately one month from discharge date.

IV. Identify demographic and clinical characteristics associated with feeling safe and unsafe.

OUTLINE:

Participants complete surveys over 15 minutes at 1-2 days before discharge and at 1 month after discharge.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are discharged from the acute cancer inpatient rehabilitation unit to personal residence (house, apartment, condominium, hotel, assisted living, etc.)
* Patients who provide informed consent
* English-speaking participants

Exclusion Criteria:

* Patients discharged to another hospital or health facility (Skilled Nursing Facility [SNF], Long Term Acute Care Hospital [LTACH], inpatient hospice, etc.)
* Patients with moderate to severe cognitive deficits as determined by speech language pathologist and/or rehabilitation physician
* Patients who were re-hospitalized at any time during study period (since completion of first survey in the hospital and discharged from the hospital until approximately one month after discharge
* Patients who were readmitted to acute inpatient rehabilitation service and previously completed both surveys

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who are discharged from the acute cancer inpatient rehabilitation unit to personal residence
Sampling Method: Non-Probability Sample
Enrollment: 261 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
Patients' perceptions regarding safety after acute inpatient rehabilitation | 1 month after discharge
  Will be assessed by Patient Continuity of Care Checklist and Perceptions Regarding Safety after Rehabilitation. At the end of study, patients' demographics and clinical characteristics will be summarized for all the patients who participated in the study by standard descriptive statistics such as mean, standard deviation, median, and range for continuous variables and frequency and proportion for categorical variables. The association between these characteristics and feeling safe will be evaluated by Wilcoxon rank sum test and chi-square (or Fisher's exact) test for continuous and categorical variables, respectively. The proportion of patients who claim they feel safe at each time will be estimated and reported along with the 95% Clopper-Pearson exact confidence interval. McNemar's test will be applied to evaluate whether the status of feeling safe has changed from the time of discharge to one month afterwards.

SECONDARY OUTCOMES:
Frequency of experiencing falls and/or near falls | 1 month after discharge
  Will be calculated and reported along with a 95% confidence interval. Furthermore, circumstances surrounding reported falls collected by question 19 and 20 in the survey will be summarized by descriptive statistics. Answers about other aspects of safety concerns collected by the questionnaire will be reported by descriptive statistics. To further investigate the association of sociodemographic and disease characteristics of patients with their perception of safety logistic regression models may be applied. Answers to "Patient Continuity of Care Checklist" questionnaire will be summarized and subscale scores will be calculated. Subscale scores will be compared between patients with different safety perception by applying Wilcoxon rank sum test. All tests will be performed two-sided and at 5% nominal significance level unless otherwise stated. Other statistical approaches may be utilized when appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Jegy Tennison, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org